CLINICAL TRIAL: NCT07209189
Title: Neoadjuvant Chemotherapy and PD-1 Inhibition for Head and Neck Cancer Treatment De-escalation (NeoScorch HN)
Brief Title: Neoadjuvant Chemotherapy and Programmed Cell Death Protein 1(PD-1) Inhibition for Head and Neck Cancer Treatment De-escalation (NeoScorch HN)
Acronym: (NeoScorch HN)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J2537; IRB00490896 (Other: The Johns Hopkins Medicine Institutional Review Board)
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma; Oral Cavity Cancer; Oropharyngeal Cancer; Laryngeal Cancer; Sinonasal Squamous Cell Carcinoma; HPV (Human Papillomavirus)-Associated Carcinoma; Skull Base Tumors; HPV 16 Positive Oropharyngeal Tumors (OPC)
Keywords: head and neck cancer; oral cancer; oropharyngeal cancer; laryngeal cancer; HPV associated; squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Papillomavirus Infections | interventions — toripalimab; Drug Therapy; Cisplatin; Carboplatin; Docetaxel; Chemoradiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Neo + Surg : Neoadjuvant Treatment and surgery (Experimental): Neoadjuvant Chemotherapy with
  * Toripalimab + Cisplatin + Docetaxel OR
  * Toripalimab + Carboplatin + Docetaxel
  Interventions: Drug: Toripalimab + Chemotherapy
- Rad+/-Chem : Adjuvant radiation or chemoradiotherapy (Experimental): Radiation or Chemotherapy will be given after the surgery
  Interventions: Radiation: Chemoradiotherapy or radiation
- Adjuvant (ADJ) treatment (Experimental): Treated with Toripalimab after adjuvant treatment
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab + Chemotherapy — Toripalimab is the study drug and will be given via IV in all arms except "Rad+/-Chem : Adjuvant radiation or chemoradiotherapy"
  Other Names: Cisplatin; Carboplatin; Docetaxel
  Arms: Neo + Surg : Neoadjuvant Treatment and surgery
Drug: Toripalimab — Study drug
  Arms: Adjuvant (ADJ) treatment
Radiation: Chemoradiotherapy or radiation — In the adjuvant phase, either radiation or chemoradiotherapy is used for treatment
  Arms: Rad+/-Chem : Adjuvant radiation or chemoradiotherapy

SUMMARY:
The NeoScorch HN study is a single institution multisite phase II trial including 3 cohorts of 25 patients each for patients with newly diagnosed locoregionally advanced, histologically confirmed, head and neck cancer eligible for curative-intent treatment, who will receive neo-adjuvant chemoimmunotherapy-based treatment as well as standard of care adjuvant treatment. The three cohorts include three different aspects of surgical de-escalation in head and neck cancer. The first cohort includes human papillomavirus independent (HPV-) squamous cell carcinoma of the head and neck. The second cohort includes HPV-associated head and neck cancer with radiographic evidence of extranodal extension in neck lymphadenopathy. The third cohort specifically includes malignancies of the sinonasal cavity and skull base which have a propensity for invasion of the orbit, skull base, and maxilla. Surgical treatment of all three of these cohorts has significant morbidity including swallowing, speech, and vision among others.

ELIGIBILITY:
Inclusion:

* Eligible subjects must have histologically confirmed, locoregionally advanced head and neck or sinonasal, nasolacrimal, or skull base tumors and meet HPV testing requirements as outlined.
* HPV-independent HNSCC (cT2-cT4, N0-N3) with potential for organ preservation using response-adapted surgery.
* HPV-associated HNSCC with radiographic extranodal extension (cT1-cT3 tonsil or lateralized base of tongue, N0-N1, up to 4 nodes with rENE).
* Sinonasal/skull base tumors, including: sinonasal carcinomas, HPV-associated sinonasal cancer, sinonasal undifferentiated carcinoma (e.g., Isocitrate dehydrogenase 2 (IDH2) mutant), or neuroendocrine sinonasal tumors (e.g., olfactory neuroblastoma) (cT2-cT4, N0-N3).
* HPV16 type only. Patients with non-HPV16 cancers are not eligible. If p16 immunohistohemistry (IHC) positivity is the only result available at enrollment, neoadjuvant therapy may start while HPV nucleic acid testing is pending. Patients found to be HPV non-16 must discontinue study participation.
* At least 8 unstained 5-µm slides must be available. If unavailable, a new biopsy is required unless waived by the PI.
* Appropriate candidates for curative-intent therapy.
* American Joint Committee on Cancer (AJCC) 7th edition: Stage III-IV, excluding N2c or bulky N2b/c (N3 equivalent) and bulky T4 (≥30cc).
* AJCC 8th edition: Stage I with N1, Stage II, or Stage III, excluding N2 disease, bulky nodal disease (N3 equivalent), or bulky T4 (≥30cc).
* Surgical arm: Candidates must be operable based on upfront imaging/exam. Patients with Grade 1 rENE may proceed to surgery; Grade 2/3 rENE are excluded.
* Measurable disease per RECIST 1.1.
* No prior systemic therapy, radiotherapy, or investigational agents for the current cancer.
* No complete surgical resection within 8 weeks of enrollment (biopsy or excision with residual disease acceptable).
* Eastern Cooperative Oncology Group (ECOG) 0-1 or Karnofsky ≥70%.
* Platelets ≥100,000/µL.
* Absolute Neutrophil Count (ANC) ≥1,500/µL.
* Hemoglobin ≥9 g/dL (without recent transfusion/EPO).
* Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) <2.5 × ULN.
* Albumin ≥2.5 mg/dL.
* Total bilirubin ≤1.5 × ULN or direct bilirubin ≤ULN if total >1.5 × ULN (Upper Limit of Normal).
* Creatinine clearance ≥60 mL/min (Cockcroft-Gault or measured GFR).
* International Normalized Ratio (INR)/ Prothrombin Time (PT) ≤1.5 × ULN (unless on anticoagulants; must be within therapeutic range).
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 × ULN (unless on anticoagulants; must be within therapeutic range).
* Must sign and understand a study-specific informed consent form.
* Women of childbearing potential (WOCBP): Negative pregnancy test within 72 hours prior to first dose.
* WOCBP must not be breastfeeding and must agree to use highly effective contraception during therapy and for 120 days after last dose.
* Men: Must use adequate contraception during treatment and for 120 days after last dose; condom use required in addition to highly effective methods.
* Azoospermic men and WOCBP not heterosexually active are exempt from contraception but must still undergo pregnancy testing.
* Counseling on pregnancy prevention is mandatory.
* Highly effective methods (<1% failure rate with consistent use) must be used

Exclusion:

* WOCBP with a positive urine pregnancy test within 72 hours before treatment allocation; if positive or inconclusive, a confirmatory serum pregnancy test is required.
* Pregnant or breastfeeding, or planning to conceive or father a child during the study and for 120 days after the last dose.
* Prior treatment with PD-1, PD-L1, PD-L2 inhibitors, or other agents targeting T-cell receptors (e.g., Cytotoxic T-lymphocyte antigen 4 (CTLA-4), OX40 (Tumor Necrosis Factor Receptor Superfamily Member 4), CD137).
* Prior systemic anti-cancer therapy or radiotherapy for the current cancer. Surgery is allowed if adequately recovered from complications.
* Radiotherapy within 2 weeks of study start. A 1-week washout is permitted for palliative, non-stereotactic radiation (≤2 weeks) to non-Central Nervous System (CNS), non-head and neck disease, provided there are no residual toxicities, no steroid requirement, and no history of radiation pneumonitis.
* Live or live-attenuated vaccines within 30 days of first study dose (including live Corona Virus Disease (COVID-19) vaccines). Inactivated, Messenger ribonucleic acid (mRNA), and peptide vaccines are allowed.
* Concurrent treatment with other investigational agents.
* Participation in another investigational drug or device study within 4 weeks before first study dose, unless in follow-up phase only.
* Diagnosis of immunodeficiency, or receiving chronic systemic steroids at doses >10 mg prednisone equivalent daily, or other immunosuppressive therapy within 7 days before study drug.
* Active autoimmune disease requiring systemic treatment in the past 2 years. Physiologic replacement therapy (thyroxine, insulin, low-dose steroids for adrenal or pituitary insufficiency) is allowed.
* History of severe hypersensitivity (≥Grade 3) to Toripalimab, its excipients, or other anti-PD-1 agents.
* Additional active malignancy requiring treatment within 2 years, except basal/squamous cell skin cancers, in situ cancers, low-grade tumors unlikely to affect survival within 3 years, or cancers treated with curative therapy.
* Active CNS metastases or carcinomatous meningitis. Intracranial extension of the primary tumor is allowed. Patients with previously treated brain metastases may enroll if radiologically stable ≥4 weeks, clinically stable, and off steroids ≥14 days before study drug.
* History of pneumonitis or interstitial lung disease requiring steroids, or current pneumonitis/Interstitial Lung Disease (ILD).
* Active infection requiring systemic therapy.
* Known HIV infection.
* Known active Hepatitis B (HBsAg positive) or active Hepatitis C (HCV RNA positive). Patients with cleared or eradicated Hepatitis B (HBV) or HCV are eligible.
* Any condition, therapy, or abnormality that could confound study results, interfere with participation, or be judged by the investigator as not in the participant's best interest.
* Known psychiatric illness or substance abuse that could interfere with study compliance. Stable chronic managed disorders are acceptable.
* History of allogeneic tissue or solid organ transplant.
* Significant cardiovascular disease, including congestive heart failure (NYHA Class III or IV), unstable angina, serious uncontrolled arrhythmia, myocardial infarction within 6 months, or prior myocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | Up to 5 years
  The objective is to achieve high-quality or "deep" responses to treatment (measurable pathologic response, MPR) that are sufficient to enable surgical de-escalation (less extensive surgery) or response-adaptive, function-preserving surgery (tailoring the surgical approach to preserve organ structure and function while maintaining oncologic safety).

CONTACTS AND LOCATIONS:
Overall Officials: Nyall R London, MD, Ph.D, Principal Investigator — Otolaryngology - Broadway

IPD SHARING:
Plan to Share IPD: No